CLINICAL TRIAL: NCT03316651
Title: A Multicenter Clinical Study of the Sequential Therapy With Whole Lung Lavage/Inhaling Granulocyte-macrophage Colony Stimulating Factor in Adult Patients With Severe Autoimmune Pulmonary Alveolar Proteinosis in China
Brief Title: Sequential Therapy With WLL/Inhaling GM-CSF for Autoimmune Pulmonary Alveolar Proteinosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dai Huaping (Other)
Responsible Party: Sponsor-Investigator, Dai Huaping, Deputy Director of Center for Respiratory Diseases, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaJapanFH001
Record Dates: First submitted 2017-08-27; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Alveolar Proteinosis; Treatment
Keywords: pulmonary alveolar proteinosis; granulocyte-macrophage colony-stimulating factor; whole lung lavage
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GM-CSF (Experimental): After the patients were randomly divided into two groups, they will receive whole lung lavage (WLL), and then one of the two groups with continue the next step as follows:
  Induction period: The time of beginning is 1 week after whole lung lavage, aerosolized GM-CSF was given for 7 days (150ug bid), and then the durg was stopped for 7 days, the 2 weeks was designed as a cycle, a total of 6 cycles (3 months) were known as the induction period.
  Maintenance period: maintenance period came up after the induction period. The dose of aerosolized GM-CSF was reduced to 150ug/d for three times a week, and then the durg was stopped for 7 days, the 2 weeks was designed as a cycle and maintenance period lasted for 9 months.
  Interventions: Drug: GM-CSF

INTERVENTIONS:
Drug: GM-CSF — After the patients were randomly divided into two groups, they will receive whole lung lavage (WLL), and then one of the two groups with continue the next step as follows:
  Induction period: The time of beginning is 1 week after whole lung lavage, aerosolized GM-CSF was given for 7 days (150ug bid), and then the durg was stopped for 7 days, the 2 weeks was designed as a cycle, a total of 6 cycles (3 months) were known as the induction period.
  Maintenance period: maintenance period came up after the induction period. The dose of aerosolized GM-CSF was reduced to 150ug/d for three times a week, and then the durg was stopped for 7 days, the 2 weeks was designed as a cycle and maintenance period lasted for 9 months.

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the sequential therapy with whole lung Lavage (WLL)/inhaling granulocyte-macrophage colony stimulating factor, compared to WLL only, for adult patients with severe autoimmune pulmonary alveolar proteinosis in China over a two-year period.

ELIGIBILITY:
Inclusion Criteria:

* Comfirmed diagnosis of autoimmune pulmonary alveolar proteinosis
* Disease severity score (DSS) is 4-5

Exclusion Criteria:

* The acute respiratory infection
* Heart failure (such as cardiogenic pulmonary edema)
* The serious liver and kidney dysfunction (creatinine or ALT were equal to or more than 2 times of the upper limit of normal range);
* Pregnancy;
* The patients with hereditary and secondary factors (inhalation of dust, hematological diseases, autoimmune diseases, etc.);
* DSS is 1-3;
* The patient is allergic to the drugs that be used in our research;
* The patients with poor compliance, or suffering from mental illness;
* The patients have not signed informed consent;
* They were treated with whole lung lavage or regular GM-CSF therapy (treatment for more than 2 weeks) within 3 months before the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to the first relapse (the date: day/month/year) | Up to 2 years
  The standard of relapse: the condition of the disease after GM-CSF inhalation meeted the standard of effective treatment or the stability criteria, and then the condition deteriorated and meeted the deteriorate standard. The standard of effective treatment: oxygenation improvement (an increase in PaO2 of more than 10mmHg and / or a reduction in A-aDO2 more than 10mmHg). The stability criteria: an increase or a reduction in PaO2 of less than 10mmHg and / a reduction or an increase in A-aDO2 of less than 10mmHg. The deteriorate standard: deteriorate oxygenation (a reduction in PaO2 of more than 10mmHg and / or an increase in A-aDO2 of more than 10mmHg).

SECONDARY OUTCOMES:
Relapse rate | Up to 2 years
FEV1 difference | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- China Japan Friendship Hispital, Beijing, China

IPD SHARING:
Plan to Share IPD: No